CLINICAL TRIAL: NCT06733740
Title: The Clinical Outcomes of Ultrasound-guided Thermal Ablation for the Treatment of Papillary Thyroid Carcinoma: A Multicenter Study
Brief Title: Ultrasound-guided Thermal Ablation for Papillary Thyroid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: 2024-655
Record Dates: First submitted 2024-12-06; First posted 2024-12-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: ultrasound-guided thermal ablation — ultrasound-guided thermal ablation to treat tumor

SUMMARY:
To evaluate long-term outcomes of ultrasound-guided thermal ablation for the treatment of papillary thyroid carcinoma

DETAILED DESCRIPTION:
To evaluate and predict long-term clinical outcomes of ultrasound-guided thermal ablation for the treatment of papillary thyroid carcinoma by a multicenter study

ELIGIBILITY:
Inclusion Criteria:

1. patients age between 18 and 80 year old, both sex
2. papillary thyroid carcinoma confirmed by core-needle biopsy or fine-needle aspiration
3. the largest diameter ≤2.0 cm
4. no clinical or imaging evidences of extrathyroidal extension, lymph node metastasis and distant metastasis on ultrasound, neck and chest CT
5. follow-up period ≥12 months

Exclusion Criteria:

1. patients with convincing evidence of aggressive papillary thyroid carcinoma or other type of thyroid cancer by biopsy
2. history of neck radiation
3. coagulation disorder, serious heart, respiratory, liver, or renal failure
4. dysfunction of the vocal cord on the opposite side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with papillary thyroid carcinoma who refuse surgery or active surveillance and choose thermal ablation
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of disease progression | through study completion, an average of 6 months
  cervical lymph node metastases, recurrent tumors and persistent tumors confirmed by pathology

SECONDARY OUTCOMES:
Rate of complications | 1 week
  complications of ablation
Rate of tumor disappearance | through study completion, an average of 6 months
  complete disappearance of ablated tumor on ultrasound and contrast-enhanced ultrasound
Rate of volume reduction | through study completion, an average of 6 months
  volume reduction of tumor after ablation on ultrasound and contrast-enhanced ultrasound
rate of change of thyroid function | through study completion, an average of 6 months
  thyroid function test, including free triiodothyronine, free thyroxine, thyroid stimulating hormone, thyroid peroxidase antibody and anti-thyroglobulin antibodies
rate of delayed surgery | through study completion, an average of 1 year
  patients underwent surgery after ablation because of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Yukun Luo, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No